CLINICAL TRIAL: NCT01234376
Title: Confocal Laser Endomicroscopy in Patients With Eosinophilic Esophagitis
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: HN-0003
Record Dates: First submitted 2010-11-02; First posted 2010-11-04 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control patients
  Interventions: Device: Confocal laser endomicroscopy
- Patients with eosinophilic esophagitis
  Interventions: Device: Confocal laser endomicroscopy

INTERVENTIONS:
Device: Confocal laser endomicroscopy — Confocal laser endomicroscopy

SUMMARY:
Confocal laser endomicroscopy enables in vivo microscopic imaging within the mucosa layer of the gut at a subcellular resolution. Various studies have addressed the potential of endomicroscopy for the in vivo diagnosis of esophageal squamous cell carcinoma, Barrett´s esophagus and esophageal adenocarcinoma. Currently, there is only one case report from our group who noted the utility of endomicroscopy for the in vivo diagnosis of eosinophilic esophagitis.

The purpose of this study is to determine whether endomicroscopy is effective for the in vivo diagnosis of eosinophilic esophagitis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 18-85 years
* Ability of subjects to understand character and individual consequences of clinical trial
* Subjects undergoing EGD

Exclusion Criteria:

* Inability to provide written informed consent
* Severe Coagulopathy (Prothrombin time < 50% of control, Partial thromboplastin time > 50 s)
* Impaired renal function (Creatinine > 1.2 mg/dl)
* Pregnancy or breast feeding
* Active gastrointestinal bleeding
* Known allergy to fluorescein, acriflavin or cresyl violet
* Residing in institutions (e.g. prison)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with eosinophilic esophagitis who underwent EGD for the evaluation of their symptoms.
  Control patients who underwent EGD because of other reasons.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Effectiveness of endomicroscopy for the in vivo diagnosis of eosinophilic esophagitis | November 2010 - November 2012

SECONDARY OUTCOMES:
Differentiation of mucosal alterations in patients with eosinophilic esophagitis compared to patients with gastroesophageal reflux disease. | November 2010 - November 2012

CONTACTS AND LOCATIONS:
Overall Officials: Markus F. Neurath, M.D., Ph.D., Study Director — University of Erlangen-Nürnberg; Helmut Neumann, M.D., Ph.D., Principal Investigator — University of Erlangen-Nürnberg
Locations (1):
- University of Erlangen-Nuremberg, Erlangen, Bavaria, Germany